CLINICAL TRIAL: NCT03668574
Title: Aerobic Exercise for Patients With Non-specific Chronic Low Back Pain: a Feasibility Randomized Controlled Trial
Brief Title: Effects of Aerobic Exercises in Patients With Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidade Cidade de Sao Paulo (Other)
Collaborators: Leonardo Oliveira Pena Costa (Unknown)
Responsible Party: Principal Investigator, Irlei dos Santos, Associate Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2.661.658
Record Dates: First submitted 2018-09-04; First posted 2018-09-12 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Low Back Pain
Keywords: Back pain; Low back pain
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise group (Experimental): Patients will firstly warm up for 5 minutes and begin training on the treadmill. There will be two weekly sessions, lasting 40 minutes, for 6 weeks, reaching a total of 12 sessions. The exercise intensity will vary from 60 to 90% of the maximum heart rate (HRmax) predicted by the percentage formula HR = HR rep + percentage (HRmax - HR rep), where HRmax = 220-age (years) and HR rep = HR obtained for five minutes of rest. Heart rate and level of subjective perception of the effort will be monitored during all sessions. Patients from this group will also be educated about their back pain by receiving a copy of The back Book.
  Interventions: Other: Aerobic exercise
- Placebo Group (Placebo Comparator): Patients will received a detuned pulsed 5-minute ultrasound and pulsed short-wave diathermy for 25 minutes, twice weekly for 6 weeks. The devices will be used with disconnected internal cables to obtain the placebo effect; however, it will be possible to manipulate the devices and adjust the doses and alarms as if they were connected, in order to simulate the pragmatism of clinical practice as well as to increase the credibility of the use of these devices in patients. Patients from this group will also be educated about their back pain by receiving a copy of The back Book.
  Interventions: Other: Placebo Group

INTERVENTIONS:
Other: Aerobic exercise — Aerobic exercise that is defined as a form of exercise lasting 15 to 60 minutes continuous and intensity of 60% to 90% of maximal heart rate.
  Arms: Aerobic exercise group
Other: Placebo Group — Will be treated with pulsed 5-minute ultrasound and pulsed short-wave diathermy for 25 minutes. The devices will be used with disconnected internal cables to obtain the placebo effect
  Arms: Placebo Group

SUMMARY:
The aim of this study is to test the feasibility of a clinical trial testing the effectiveness of aerobic exercises program in patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
A total of 30 patients with chronic non-specific low back pain (with a duration of at least 12 weeks) who are seeking for treatment will be recruited. These patients will be randomly allocated into two groups.

Patients allocated to the placebo group will be treated twice a week for a total of 12 weeks with detuned ultrasound and shortwave therapy

Patients allocated to the exercise group will be trained with aerobic exercises on a treadmill twice a week for a total of 12 weeks.

Primary outcomes will be pain and disability. Feasibility outcomes will be adherence, satisfaction and recruitment. Kinesiophobia, perceived global effect and physical capacity will also be analyzed as secondary outcomes. The outcome assessor of this trial will be blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic non-specific low back pain with a pain intensity of at least 3 points at the baseline assessment measured by the Numerical Pain Scale, between 18 and 80 years of age and able to read Portuguese.

Exclusion Criteria:

* Patients who have some contraindication to exercise, fractures, tumors, inflammatory and infectious diseases, severe cardiovascular and metabolic diseases, and the development of chronic inflammatory diseases (eg, dyspnoea, limiting diseases of the lower limbs, previous spinal surgery and pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measured by a 0-10 Numerical Pain Rating Scale. | Six weeks after randomization
  Pain intensity will be measured by a 0-10 Numerical Pain Rating Scale. Higher values represent higher pain intensity.

SECONDARY OUTCOMES:
Disability measured with the 0-24 Rolland Morris Disability Questionnaire. | Six weeks after randomization
  Disability will be measured with the 0-24 Rolland Morris Disability Questionnaire. Higher values represent higher disability.
Kinesiophobia measured with Tampa Scale of Kinesiophobia | Six weeks after randomization
  Kinesiophobia (i.e. fear of movement) will be measured with the 17-68 point Tampa Scale of kinesiophobia. The higher the score, the higher is the fear of movement.
Global Impression of Recovery measured with the 11-point Global Perceived Effect Scale | Six weeks after randomization
  Global impression of recovery will be measured with the 11-point (-5 to + 5) Global Perceived Effect Scale. A negative score means deterioration of symptoms and positive scores mean improvement. A score of +5 means that the patient is considered as fully recovered.
Physical activity levels measured with an Accelerometer | Six weeks after randomization
  Physical Activity will be measured with an accelerometer. Patients will wear an accelerometer for seven consecutive days. The higher the values, the higher the physical activity levels.
Maximum exercise capacity measured with the modified Shuttle Walk Test | Six weeks after randomization
  Maximum exercise capacity will be measured with the modified Shuttle Walk Test. The purpose of this test is to see how far and fast patients can walk by following a series of time signals.
  Patients will be asked to walk between two cones spaced 10 metres apart. Participants will begin by walking at a very slow pace; this pace is set by a beep. Patients will walk around the 10 metre course aiming to turn around a cone at the first beep, and around the second cone at the next beep.
  The beep's will very gradually get faster, which means that patients will begin to walk at a quicker pace, getting faster and faster until he/she cannot keep up with the set pace, or until the participant is too breathless or tired to continue.
  The test has 12 levels each lasting 1 minute with a minimum walking speed of 1.2 miles per hour, up to a maximum of 5.3 miles per hour.

OTHER OUTCOMES:
Adherence | Six weeks after randomization
  This is the first measure to test if a larger trial will be feasible: the investigators will count the number of treatment sessions that patients attended during the treatment phase of the trial. The higher the number, the higher the adherence.
Recruitment measures | Prior to randomisation
  The investigators will record the number of patients who will not agree to participate in the study and reasons for declining.
Satisfaction with care measured with the 0-130 Medrisk Patient Satisfaction Questionnaire | Six weeks after randomization
  The investigators will use the 0-130 Medrisk Patient Satisfaction Questionnaire for measuring satisfaction with care. The higher the score, the higher is the satisfaction with care.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Costa, PhD, Principal Investigator — Universidade Cidade de Sao Paulo
Locations (1):
- Irlei dos Santos, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] van der Velde G, Mierau D. The effect of exercise on percentile rank aerobic capacity, pain, and self-rated disability in patients with chronic low-back pain: a retrospective chart review. Arch Phys Med Rehabil. 2000 Nov;81(11):1457-63. doi: 10.1053/apmr.2000.9629. PMID 11083348
- [Background] Stochkendahl MJ, Kjaer P, Hartvigsen J, Kongsted A, Aaboe J, Andersen M, Andersen MO, Fournier G, Hojgaard B, Jensen MB, Jensen LD, Karbo T, Kirkeskov L, Melbye M, Morsel-Carlsen L, Nordsteen J, Palsson TS, Rasti Z, Silbye PF, Steiness MZ, Tarp S, Vaagholt M. National Clinical Guidelines for non-surgical treatment of patients with recent onset low back pain or lumbar radiculopathy. Eur Spine J. 2018 Jan;27(1):60-75. doi: 10.1007/s00586-017-5099-2. Epub 2017 Apr 20. PMID 28429142
- [Background] Meng XG, Yue SW. Efficacy of aerobic exercise for treatment of chronic low back pain: a meta-analysis. Am J Phys Med Rehabil. 2015 May;94(5):358-65. doi: 10.1097/PHM.0000000000000188. PMID 25299528
- [Background] Chiarotto A, Boers M, Deyo RA, Buchbinder R, Corbin TP, Costa LOP, Foster NE, Grotle M, Koes BW, Kovacs FM, Lin CC, Maher CG, Pearson AM, Peul WC, Schoene ML, Turk DC, van Tulder MW, Terwee CB, Ostelo RW. Core outcome measurement instruments for clinical trials in nonspecific low back pain. Pain. 2018 Mar;159(3):481-495. doi: 10.1097/j.pain.0000000000001117. PMID 29194127
- [Background] de Fatima Costa Oliveira N, Oliveira Pena Costa L, Nelson R, Maher CG, Beattie PF, de Bie R, Oliveira W, Camara Azevedo D, da Cunha Menezes Costa L. Measurement properties of the Brazilian Portuguese version of the MedRisk instrument for measuring patient satisfaction with physical therapy care. J Orthop Sports Phys Ther. 2014 Nov;44(11):879-89. doi: 10.2519/jospt.2014.5150. PMID 25361861
- [Background] Gordon R, Bloxham S. A Systematic Review of the Effects of Exercise and Physical Activity on Non-Specific Chronic Low Back Pain. Healthcare (Basel). 2016 Apr 25;4(2):22. doi: 10.3390/healthcare4020022. PMID 27417610